CLINICAL TRIAL: NCT04442490
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Efficacy of SAGE-217 in the Treatment of Adult Subjects With Major Depressive Disorder
Brief Title: A Study to Evaluate the Efficacy of Sage-217 in the Treatment of Adult Participants With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-MDD-301B
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Depressive disorder; SAGE-217
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants self-administered SAGE-217 matched-placebo capsules, once daily at approximately 8 PM with fat-containing food for 14 days.
  Interventions: Drug: Placebo
- SAGE-217 50 mg (Experimental): Participants self-administered SAGE-217 50 mg capsules, once daily at approximately 8 PM with fat-containing food for 14 days. Participants who could not tolerate 50 mg received 40 mg for the remainder of the treatment period as per discretion of investigator.
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217 oral capsules.
  Arms: SAGE-217 50 mg
Drug: Placebo — SAGE-217 matched-placebo oral capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study to evaluate the efficacy of SAGE-217 in the treatment of participants with MDD.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant with diagnosis of MDD as diagnosed by Structured Clinical Interview for Diagnostic and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Clinical Trial Version [SCID-5-CT], with symptoms that have been present for at least a 4-week period.
2. Participant has a Hamilton Rating Scale for Depression (HAM-D) total score ≥24 at screening and Day 1 (prior to dosing).
3. Participants taking antidepressants must have been taking these medications at the same dose for at least 60 days prior to Day 1. Participants who have stopped taking antidepressants within 60 days must have stopped for longer than 5 half-lives of the antidepressant prior to Day 1. Participants receiving psychotherapy must have been receiving therapy on a regular schedule for at least 60 days prior to Day 1.
4. Participant is willing to delay start of other antidepressant or antianxiety medications and any new pharmacotherapy regimens, including as-needed benzodiazepine anxiolytics and sleep aids, until after completion of the Day 42 visit.

Exclusion Criteria:

1. Participant is currently at significant risk of suicide, as judged by the Investigator, or has attempted suicide associated with the current episode of MDD.
2. Participant has onset of the current depressive episode during pregnancy or 4 weeks postpartum, or the participant has presented for screening during the 6-month postpartum period.
3. Participant has a body mass index (BMI) ≤18 or ≥45 kg/m^2 at Screening, which is subject to a broader evaluation of medical comorbidities.
4. Participant has treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants within the current major depressive episode (excluding antipsychotics) from two different classes for at least 4 weeks of treatment.
5. Participant has a medical history of seizures, bipolar disorder, schizophrenia, and/or schizoaffective disorder.
6. Participant has a history of mild, moderate, or severe substance use disorder (including benzodiazepines) diagnosed using DSM-5 criteria in the 12 months prior to screening.
7. Participant is taking psychostimulants (eg, methylphenidate, amphetamine) or opioids, regularly or as-needed, at Day -28.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 543 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Bellflower, California
  - Sage Investigational Site, Garden Grove, California
  - Sage Investigational Site, Glendale, California
  - Sage Investigational Site, Lemon Grove, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Pico Rivera, California
  - Sage Investigational Site, Redlands, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Sherman Oaks, California
  - Sage Investigational Site, Temecula, California
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Lauderhill, Florida
  - Sage Investigational Site, Orange City, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Alpharetta, Georgia
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Skokie, Illinois
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, O'Fallon, Missouri
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Marlton, New Jersey
  - Sage Investigational Site, Charlotte, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, North Canton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Portland, Oregon
  - Sage Investigational Site, Allentown, Pennsylvania
  - Sage Investigational Site, Charleston, South Carolina
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, DeSoto, Texas
  - Sage Investigational Site, Wichita Falls, Texas
  - Sage Investigational Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 39 centers in the United States from 12 May 2020 to 21 April 2021.
Pre-assignment Details: A total of 543 participants were randomized, of which 543 were enrolled in this study and 537 received Investigational Product (IP). Part B was started after all participants in Part A (NCT03672175) completed Day 42 of the previous study.
Groups:
- SAGE-217 50 mg: Participants self-administered SAGE-217 50 mg capsules, once daily at approximately 8 PM with fat-containing food for 14 days. Participants who could not tolerate 50 milligrams (mg) received 40 mg for the remainder of the treatment period as per discretion of investigator.
Period: Overall Study
Arm/Group | Placebo | SAGE-217 50 mg
Started | 272 | 271
Safety Set (Safety Set included all participants who were administered investigational product (IP).) | 269 | 268
Completed | 235 | 242
Not Completed | 37 | 29
Not completed — Withdrawal by Subject | 18 | 10
Not completed — Lost to Follow-up | 7 | 7
Not completed — Adverse Event | 2 | 6
Not completed — Noncompliance | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Reason not Specified | 2 | 1
Not completed — Randomized but not Treated | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-217 50 mg | Total
Number analyzed (Participants) | 269 | 268 | 537
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.64) | 39.4 (12.30) | 39.7 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 186 | 352
  Male | 103 | 82 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 58 | 112
  Not Hispanic or Latino | 215 | 210 | 425
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 4 | 13 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 46 | 75 | 121
  White | 206 | 169 | 375
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 4 | 2 | 6
17-item Hamilton Rating Scale for Depression (HAM-D) Total Score [Mean (Standard Deviation); unit: score on a scale] — The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total HAM-D score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression.
  score on a scale | 26.9 (2.67) | 26.8 (2.60) | 26.9 (2.64)
Clinical Global Impression - Severity (CGIS) Score [Mean (Standard Deviation); unit: score on a scale] — The CGI-S is a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. A participant is assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7= among the most extremely ill participants
  score on a scale | 4.8 (0.52) | 4.7 (0.55) | 4.7 (0.54)
Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. The MADRS total score was calculated as the sum of the 10 individual item scores and each item yields a score of 0 to 6. The total MADRS score ranges from 0 to 60, where higher scores indicate more severe depression.
  score on a scale | 35.0 (4.73) | 35.2 (4.83) | 35.1 (4.78)
Hamilton Anxiety Rating Scale (HAM-A) Total Score [Mean (Standard Deviation); unit: score on a scale] — The 14-item HAM-A is comprised of a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The HAM-A total score will be calculated as the sum of the 14 individual item scores. The scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe) with a total HAM-A score range of 0 to 56, where less than (<)17 indicates mild severity, 18 to 24 indicates mild to moderate severity, and 25 to 30 indicates moderate to severe severity. Population: "Number analyzed" = Number of participants evaluable for the specified baseline measure.
  score on a scale
    number analyzed (Participants) | 268 | 268 | 536
    (all) | 20.7 (5.51) | 21.4 (5.15) | 21.0 (5.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 17-item HAM-D Total Score at Day 15
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total HAM-D score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression. A negative change indicates improvement. A mixed Model for Repeated Measures (MMRM)was used for the analysis.
Time Frame: Baseline, Day 15
Population: The FAS included all randomized participants who were administered IP with valid baseline HAM-D total score and had at least 1 valid post-baseline HAM-D total score. Overall number of participants analyzed are the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 251 | 248
score on a scale | -12.3 (0.50) | -14.1 (0.51)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Test type: Superiority; p = 0.0141, MMRM; Least Squares (LS) Mean Difference = -1.7, 95% CI 2-sided [-3.1 to -0.3], Standard Error of Mean 0.70 — Model used was the MMRM with treatment, baseline HAM-D total score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction as fixed effects with Unstructured covariance structure

2. Secondary Outcome: Change From Baseline in the CGI-S Score at Day 15
Description: The CGI-S is a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. A participant is assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7= among the most extremely ill participants. A negative change from baseline indicates improvement. MMRM was used for the analysis. A negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Day 15
Population: FAS included all randomized participants who were administered IP with valid baseline HAM-D total score and had at least 1 valid post-baseline HAM-D total score. Overall number of participants analyzed are the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 268 | 266
score on a scale | -1.6 (0.08) | -1.8 (0.08)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Test type: Superiority; p = 0.1193, MMRM; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.11 — Model used was the MMRM with treatment (SAGE-217 or placebo), baseline CGI-S score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction as fixed effects with Unstructured covariance structure

3. Secondary Outcome: Change From Baseline in the HAM-D Total Score at Days 3, 8 and 42
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total HAM-D score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression. A negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 3, 8, and 42
Population: FAS included all randomized participants who were administered IP with valid baseline HAM-D total score and had at least 1 valid post-baseline HAM-D total score. Number analyzed is the number of participants with data available for analysis at the given timepoints.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 268 | 266
score on a scale
  Change from Baseline at Day 3: number analyzed (Participants) | 264 | 263
  Change from Baseline at Day 3 | -6.8 (0.38) | -9.8 (0.38)
  Change from Baseline at Day 8: number analyzed (Participants) | 262 | 255
  Change from Baseline at Day 8 | -9.5 (0.45) | -12.0 (0.45)
  Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Change from Baseline at Day 42 | -12.6 (0.55) | -13.5 (0.55)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from baseline at Day 3; Test type: Superiority; p < 0.0001, MMRM; LS Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -2.0], Standard Error of Mean 0.52 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Change from baseline at Day 8; Test type: Superiority; p < 0.0001, MMRM; LS Mean Difference = -2.6, 95% CI 2-sided [-3.8 to -1.4], Standard Error of Mean 0.61 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SAGE-217 50 mg; Change from baseline at Day 42; Test type: Superiority; p = 0.2344, MMRM; LS Mean Difference = -0.9, 95% CI 2-sided [-2.4 to 0.6], Standard Error of Mean 0.76 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving HAM-D Response
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total HAM-D score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression. HAM-D response is defined as having a greater than or equal to (≥) 50% reduction in HAM-D score from baseline. Generalized Estimating Equation (GEE) method was used for the analysis.
Time Frame: Days 15 and 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 268 | 266
percentage of participants
  Day 15: number analyzed (Participants) | 251 | 248
  Day 15 | 47.0 | 56.0
  Day 42: number analyzed (Participants) | 233 | 240
  Day 42 | 45.9 | 52.9
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Day 15; Test type: Superiority; p = 0.0599, Generalized Estimating Equation Model; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.99 to 1.98]; Model used is a GEE for binary response model, with factors for treatment, baseline HAM-D total score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction with Unstructured covariance structure. Odds ratio was the estimate of the odds of having HAM-D response for participants treated with SAGE-217 relative to that for participants treated with placebo
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Day 42; Test type: Superiority; p = 0.0889, GEE Model; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.94]; Model used is a GEE for binary response model, with factors for treatment, baseline HAM-D total score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction with Unstructured covariance structure.Odds ratio was the estimate of the odds of having HAM-D response for participants treated with SAGE-217 relative to that for participants treated with placebo

5. Secondary Outcome: Percentage of Participants Achieving HAM-D Remission
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to the following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total HAM-D score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression. HAM-D remission is defined as HAM-D total score less than or equal to (≤) 7. GEE model was used for the analysis.
Time Frame: Days 15 and 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 268 | 266
percentage of participants
  Day 15: number analyzed (Participants) | 251 | 248
  Day 15 | 27.1 | 29.8
  Day 42: number analyzed (Participants) | 233 | 240
  Day 42 | 29.6 | 30.8
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Day 15; Test type: Superiority; p = 0.5495, GEE Model; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.76 to 1.66]; Model used is GEE for binary response model, with factors for treatment, baseline HAM-D total score, antidepressant use at baseline, assessment time point, and time point-by-treatment interaction with Unstructured covariance structure. Odds ratio was the estimate of the odds of having HAM-D remission for participants treated with SAGE-217 relative to that for participants treated with placebo
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Day 42; Test type: Superiority; p = 0.6790, GEE Model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.74 to 1.60]; [other analysis details as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response at Day 15
Description: CGI-I response is defined as having a CGI-I score of "very much improved" (score of 1) or "much improved" (score of 2)". The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. Response choices include 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. GEE model was used for the analysis.
Time Frame: Day 15
Population: FAS included all randomized participants who were administered IP with valid baseline HAM-D total score and had at least 1 valid post-baseline HAM-D total score. Overall number of participants is the participants with response.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 251 | 248
percentage of participants | 51.0 | 62.1
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Placebo, SAGE-217; Test type: Superiority; p = 0.0191, GEE Model; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.07 to 2.16]; Model used was a GEE for binary response model, with factors for treatment, CGI-S baseline score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction with Unstructured covariance structure. Odds ratio was the estimate of the odds of having CGI-I response for participants treated with SAGE-217 relative to that for participants treated with placebo

7. Secondary Outcome: Change From Baseline in MADRS Total Score at Day 15
Description: The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. The MADRS total score was calculated as the sum of the 10 individual item scores and each item yields a score of 0 to 6. The overall MADRS score ranges from 0 to 60 where higher MADRS scores indicate more severe depression. A negative change indicates improvement. MMRM was used analysis.
Time Frame: Baseline, Day 15
Population: FAS included all randomized participants who were administered IP with valid baseline HAM-D total score and had at least 1 valid post-baseline HAM-D total score. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 251 | 247
score on a scale | -15.1 (0.76) | -17.5 (0.77)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Placebo, SAGE-217; Test type: Superiority; p = 0.0238, MMRM; LS Mean Difference = -2.4, 95% CI 2-sided [-4.4 to -0.3], Standard Error of Mean 1.05 — Model used was the MMRM with treatment (SAGE-217/placebo), baseline MADRS total score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction as fixed effects with Unstructured covariance structure

8. Secondary Outcome: Change From Baseline in HAM-A Total Score at Day 15
Description: The 14-item HAM-A is comprised of a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The HAM-A total score was calculated as the sum of the 14 individual item scores. The scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe) to each item, with a total HAM-A score range of 0 to 56, where <17 indicates mild severity, 18 to 24 indicates mild to moderate severity, and 25 to 30 indicates moderate to severe severity. A negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Day 15
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 251 | 247
score on a scale | -9.1 (0.43) | -10.4 (0.43)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Placebo, SAGE-217; Test type: Superiority; p = 0.0199, MMRM; LS Mean Difference = -1.4, 95% CI 2-sided [-2.5 to -0.2], Standard Error of Mean 0.58 — Model used was MMRM with treatment (SAGE-217/placebo), baseline HAM-A total score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction as fixed effects with Unstructured covariance structure

9. Secondary Outcome: Time to First HAM-D Response
Description: 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. Total HAM-D score is sum of individual items, ranging from 0 to 52; where higher score indicates more depression. Time to first HAM-D response is defined as time from first administration of the study drug to first time when ≥50% reduction in HAM-D score from baseline is achieved.
Time Frame: Up to Day 57
Population: FAS included all randomized participants who were administered IP with valid baseline HAM-D total score and had at least 1 valid post-baseline HAM-D total score. Overall number of participants analyzed is the number of participants with response.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 166 | 197
days | 15 [2 to 57] | 11 [2 to 54]

10. Secondary Outcome: Change From Baseline in Patient- Reported Outcome (PRO) Measures of Health-Related Quality of Life, as Assessed by the 36-item Short Form Version 2 (SF-36v2) Score at Days 8, 15, 28 and 42
Description: Participant's health was assessed using PRO health related quality of life (HRQOL) SF-36 V2. SF-36v2 covers 8 health dimensions, including 4 physical health status domains (physical functioning, role participation with physical health problems [role-physical], bodily pain, and general health) and 4 mental health status domains (vitality, social functioning, role participation with emotional health problems [role-emotional], and mental health). Physical Component Summary and the Mental Component Summary are derived from the 8 domains. Each domain is scored by summing the individual items, scores varying between 0 and 100. Both the domain scores and the component summary scores are norm-based. A higher score indicates a better state of health. Positive change indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 8, 15, 28 and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 268 | 266
score on a scale
  Physical Functioning Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Physical Functioning Domain Score: Change from Baseline at Day 8 | 1.9 (0.36) | 2.4 (0.37)
  Physical Functioning Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Physical Functioning Domain Score: Change from Baseline at Day 15 | 2.3 (0.38) | 3.1 (0.39)
  Physical Functioning Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Physical Functioning Domain Score: Change from Baseline at Day 28 | 2.3 (0.40) | 3.2 (0.41)
  Physical Functioning Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Physical Functioning Domain Score: Change from Baseline at Day 42 | 2.4 (0.43) | 3.3 (0.43)
  Role-Physical Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Role-Physical Domain Score: Change from Baseline at Day 8 | 1.9 (0.43) | 1.8 (0.44)
  Role-Physical Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Role-Physical Domain Score: Change from Baseline at Day 15 | 3.2 (0.45) | 3.1 (0.46)
  Role-Physical Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Role-Physical Domain Score: Change from Baseline at Day 28 | 3.1 (0.46) | 3.0 (0.46)
  Role-Physical Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Role-Physical Domain Score: Change from Baseline at Day 42 | 3.2 (0.46) | 3.5 (0.46)
  Bodily Pain Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Bodily Pain Domain Score: Change from Baseline at Day 8 | 3.3 (0.46) | 3.8 (0.47)
  Bodily Pain Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Bodily Pain Domain Score: Change from Baseline at Day 15 | 4.7 (0.49) | 4.9 (0.50)
  Bodily Pain Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Bodily Pain Domain Score: Change from Baseline at Day 28 | 4.7 (0.51) | 5.0 (0.51)
  Bodily Pain Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Bodily Pain Domain Score: Change from Baseline at Day 42 | 4.2 (0.54) | 5.2 (0.54)
  General Health Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  General Health Domain Score: Change from Baseline at Day 8 | 2.4 (0.36) | 3.6 (0.37)
  General Health Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  General Health Domain Score: Change from Baseline at Day 15 | 3.4 (0.39) | 4.4 (0.40)
  General Health Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  General Health Domain Score: Change from Baseline at Day 28 | 3.3 (0.43) | 3.8 (0.43)
  General Health Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  General Health Domain Score: Change from Baseline at Day 42 | 3.5 (0.45) | 4.6 (0.45)
  Vitality Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Vitality Domain Score: Change from Baseline at Day 8 | 7.2 (0.64) | 9.8 (0.65)
  Vitality Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Vitality Domain Score: Change from Baseline at Day 15 | 9.7 (0.75) | 12.8 (0.76)
  Vitality Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Vitality Domain Score: Change from Baseline at Day 28 | 9.1 (0.75) | 10.9 (0.76)
  Vitality Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Vitality Domain Score: Change from Baseline at Day 42 | 9.7 (0.81) | 11.7 (0.81)
  Social Functioning Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Social Functioning Domain Score: Change from Baseline at Day 8 | 8.2 (0.66) | 9.5 (0.67)
  Social Functioning Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Social Functioning Domain Score: Change from Baseline at Day 15 | 11.4 (0.72) | 12.5 (0.73)
  Social Functioning Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Social Functioning Domain Score: Change from Baseline at Day 28 | 11.6 (0.76) | 11.9 (0.76)
  Social Functioning Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Social Functioning Domain Score: Change from Baseline at Day 42 | 11.4 (0.78) | 13.2 (0.78)
  Role-Emotional Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Role-Emotional Domain Score: Change from Baseline at Day 8 | 9.4 (0.77) | 10.5 (0.78)
  Role-Emotional Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Role-Emotional Domain Score: Change from Baseline at Day 15 | 12.1 (0.82) | 13.6 (0.83)
  Role-Emotional Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Role-Emotional Domain Score: Change from Baseline at Day 28 | 11.8 (0.84) | 13.7 (0.84)
  Role-Emotional Domain Score: Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Role-Emotional Domain Score: Change from Baseline at Day 42 | 12.3 (0.89) | 13.5 (0.89)
  Mental Health Domain Score: Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Mental Health Domain Score: Change from Baseline at Day 8 | 9.4 (0.68) | 11.0 (0.69)
  Mental Health Domain Score: Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Mental Health Domain Score: Change from Baseline at Day 15 | 12.2 (0.76) | 14.0 (0.77)
  Mental Health Domain Score: Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Mental Health Domain Score: Change from Baseline at Day 28 | 11.6 (0.81) | 12.7 (0.81)
  Mental Health Domain Score: Change from Baseline at Day 42 | 12.2 (0.85) | 13.9 (0.85)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Physical Functioning Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.3216, MMRM; LS Mean Difference = 0.5, 95% CI 2-sided [-0.5 to 1.5], Standard Error of Mean 0.50 — Model used is MMRM with treatment(SAGE-217/placebo), baseline SF-36v2 domain/component score, antidepressant use at baseline(Yes/No)assessment time point and time point-by-treatment interaction as fixed effects with Unstructured covariance structure
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Physical Functioning Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.1247, MMRM; LS Mean Difference = 0.8, 95% CI 2-sided [-0.2 to 1.8], Standard Error of Mean 0.53 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SAGE-217 50 mg; Physical Functioning Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.1111, MMRM; LS Mean Difference = 0.9, 95% CI 2-sided [-0.2 to 2.0], Standard Error of Mean 0.56 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SAGE-217 50 mg; Physical Functioning Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.1449, MMRM; LS Mean Difference = 0.9, 95% CI 2-sided [-0.3 to 2.0], Standard Error of Mean 0.59 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SAGE-217 50 mg; Role-Physical Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.8242, MMRM; LS Mean Difference = -0.1, 95% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.59 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SAGE-217 50 mg; Role-Physical Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.8329, MMRM; LS Mean Difference = -0.1, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.62
Statistical Analysis 7: Comparison: Placebo vs SAGE-217 50 mg; Role-Physical Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.8127, MMRM; LS Mean Difference = -0.1, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.63
Statistical Analysis 8: Comparison: Placebo vs SAGE-217 50 mg; Role-Physical Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.5435, MMRM; LS Mean Difference = 0.4, 95% CI 2-sided [-0.9 to 1.6], Standard Error of Mean 0.64
Statistical Analysis 9: Comparison: Placebo vs SAGE-217 50 mg; Bodily Pain Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.3551, MMRM; LS Mean Difference = 0.6, 95% CI 2-sided [-0.7 to 1.8], Standard Error of Mean 0.63
Statistical Analysis 10: Comparison: Placebo vs SAGE-217 50 mg; Bodily Pain Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.7495, MMRM; LS Mean Difference = 0.2, 95% CI 2-sided [-1.1 to 1.6], Standard Error of Mean 0.68
Statistical Analysis 11: Comparison: Placebo vs SAGE-217 50 mg; Bodily Pain Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.6471, MMRM; LS Mean Difference = 0.3, 95% CI 2-sided [-1.1 to 1.7], Standard Error of Mean 0.70
Statistical Analysis 12: Comparison: Placebo vs SAGE-217 50 mg; Bodily Pain Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.1832, MMRM; LS Mean Difference = 1.0, 95% CI 2-sided [-0.5 to 2.5], Standard Error of Mean 0.75
Statistical Analysis 13: Comparison: Placebo vs SAGE-217 50 mg; General Health Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.0168, MMRM; LS Mean Difference = 1.2, 95% CI 2-sided [0.2 to 2.2], Standard Error of Mean 0.50
Statistical Analysis 14: Comparison: Placebo vs SAGE-217 50 mg; General Health Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.0787, MMRM; LS Mean Difference = 1.0, 95% CI 2-sided [-0.1 to 2.0], Standard Error of Mean 0.54
Statistical Analysis 15: Comparison: Placebo vs SAGE-217 50 mg; General Health Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.4273, MMRM; LS Mean Difference = 0.5, 95% CI 2-sided [-0.7 to 1.6], Standard Error of Mean 0.59
Statistical Analysis 16: Comparison: Placebo vs SAGE-217 50 mg; General Health Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.0938, MMRM; LS Mean Difference = 1.0, 95% CI 2-sided [-0.2 to 2.2], Standard Error of Mean 0.62
Statistical Analysis 17: Comparison: Placebo vs SAGE-217 50 mg; Vitality Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.0033, MMRM; LS Mean Difference = 2.6, 95% CI 2-sided [0.9 to 4.3], Standard Error of Mean 0.88
Statistical Analysis 18: Comparison: Placebo vs SAGE-217 50 mg; Vitality Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.0029, MMRM; LS Mean Difference = 3.1, 95% CI 2-sided [1.1 to 5.1], Standard Error of Mean 1.03
Statistical Analysis 19: Comparison: Placebo vs SAGE-217 50 mg; Vitality Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.0791, MMRM; LS Mean Difference = 1.8, 95% CI 2-sided [-0.2 to 3.9], Standard Error of Mean 1.04
Statistical Analysis 20: Comparison: Placebo vs SAGE-217 50 mg; Vitality Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.0761, MMRM; LS Mean Difference = 2.0, 95% CI 2-sided [-0.2 to 4.2], Standard Error of Mean 1.12
Statistical Analysis 21: Comparison: Placebo vs SAGE-217 50 mg; Social Functioning Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.1568, MMRM; LS Mean Difference = 1.3, 95% CI 2-sided [-0.5 to 3.1], Standard Error of Mean 0.91
Statistical Analysis 22: Comparison: Placebo vs SAGE-217 50 mg; Social Functioning Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.2807, MMRM; LS Mean Difference = 1.1, 95% CI 2-sided [-0.9 to 3.0], Standard Error of Mean 0.99
Statistical Analysis 23: Comparison: Placebo vs SAGE-217 50 mg; Social Functioning Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.7751, MMRM; LS Mean Difference = 0.3, 95% CI 2-sided [-1.8 to 2.4], Standard Error of Mean 1.05
Statistical Analysis 24: Comparison: Placebo vs SAGE-217 50 mg; Social Functioning Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.0913, MMRM; LS Mean Difference = 1.8, 95% CI 2-sided [-0.3 to 3.9], Standard Error of Mean 1.07
Statistical Analysis 25: Comparison: Placebo vs SAGE-217 50 mg; Role-Emotional Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.2863, MMRM; LS Mean Difference = 1.1, 95% CI 2-sided [-0.9 to 3.2], Standard Error of Mean 1.05
Statistical Analysis 26: Comparison: Placebo vs SAGE-217 50 mg; Role-Emotional Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.1801, MMRM; LS Mean Difference = 1.5, 95% CI 2-sided [-0.7 to 3.7], Standard Error of Mean 1.13
Statistical Analysis 27: Comparison: Placebo vs SAGE-217 50 mg; Role-Emotional Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.1107, MMRM; LS Mean Difference = 1.8, 95% CI 2-sided [-0.4 to 4.1], Standard Error of Mean 1.16
Statistical Analysis 28: Comparison: Placebo vs SAGE-217 50 mg; Role-Emotional Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.3274, MMRM; LS Mean Difference = 1.2, 95% CI 2-sided [-1.2 to 3.6], Standard Error of Mean 1.23
Statistical Analysis 29: Comparison: Placebo vs SAGE-217 50 mg; Mental Health Domain Score: Change from Baseline at Day 8; Test type: Superiority; p = 0.0873, MMRM; LS Mean Difference = 1.6, 95% CI 2-sided [-0.2 to 3.4], Standard Error of Mean 0.93
Statistical Analysis 30: Comparison: Placebo vs SAGE-217 50 mg; Mental Health Domain Score: Change from Baseline at Day 15; Test type: Superiority; p = 0.0871, MMRM; LS Mean Difference = 1.8, 95% CI 2-sided [-0.3 to 3.9], Standard Error of Mean 1.05
Statistical Analysis 31: Comparison: Placebo vs SAGE-217 50 mg; Mental Health Domain Score: Change from Baseline at Day 28; Test type: Superiority; p = 0.3095, MMRM; LS Mean Difference = 1.1, 95% CI 2-sided [-1.1 to 3.3], Standard Error of Mean 1.12
Statistical Analysis 32: Comparison: Placebo vs SAGE-217 50 mg; Mental Health Domain Score: Change from Baseline at Day 42; Test type: Superiority; p = 0.1477, MMRM; LS Mean Difference = 1.7, 95% CI 2-sided [-0.6 to 4.0], Standard Error of Mean 1.17

11. Secondary Outcome: Change From Baseline in PRO Measures of Depressive Symptoms, as Assessed by the 9-item Patient Health Questionnaire (PHQ-9) Total Score at Days 8, 15, 28 and 42
Description: The PHQ-9 is a participant-rated depressive symptom severity scale where scoring is based on responses to specific questions. The score was calculated as the sum of the 9 individual item scores. The PHQ-9 total score ranges from 0 to 27 categorized as follows: 1 to 4 = minimal depression, 5 to 9 = mild depression, 10 to 14 = moderate depression, 15 to 19 = moderately severe depression, and 20 to 27 = severe depression with a higher score indicating more depression. A negative change indicates improvements. MMRM was used for analysis.
Time Frame: Baseline, Days 8, 15, 28 and 42
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 268 | 266
score on a scale
  Change from Baseline at Day 8: number analyzed (Participants) | 261 | 255
  Change from Baseline at Day 8 | -6.8 (0.42) | -7.8 (0.42)
  Change from Baseline at Day 15: number analyzed (Participants) | 251 | 247
  Change from Baseline at Day 15 | -8.3 (0.45) | -9.4 (0.46)
  Change from Baseline at Day 28: number analyzed (Participants) | 233 | 237
  Change from Baseline at Day 28 | -7.8 (0.46) | -8.8 (0.46)
  Change from Baseline at Day 42: number analyzed (Participants) | 233 | 240
  Change from Baseline at Day 42 | -8.5 (0.48) | -9.0 (0.48)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 8; Test type: Superiority; p = 0.0828, MMRM; LS Mean Difference = -1.0, 95% CI 2-sided [-2.1 to 0.1], Standard Error of Mean 0.57 — Model used was the MMRM with treatment (SAGE-217/placebo), baseline PHQ-9 total score, antidepressant use at baseline (Yes or No), assessment time point, and time point-by-treatment interaction as fixed effects with Unstructured covariance structure
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.0606, MMRM; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.62 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 28; Test type: Superiority; p = 0.1079, MMRM; LS Mean Difference = -1.0, 95% CI 2-sided [-2.3 to 0.2], Standard Error of Mean 0.63 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 42; Test type: Superiority; p = 0.3951, MMRM; LS Mean Difference = -0.6, 95% CI 2-sided [-1.9 to 0.7], Standard Error of Mean 0.66 — [estimate comment as in outcome 11, analysis 1]

ADVERSE EVENTS:
Time Frame: From inform consent signing up to 28 days after the last dose (Up to 70 days)
Description: Safety set included all participants who were administered IP.
Arm/Group | Placebo | SAGE-217 50 mg
All-Cause Mortality (participants affected / at risk) | 0/269 | 0/268
Serious Adverse Events (participants affected / at risk) | 2/269 | 2/268
Other Adverse Events (participants affected / at risk) | 59/269 | 111/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=269) | SAGE-217 50 mg (N=268)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Slow Speech (Nervous system disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Gamma-glutamyltransferase Increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=269) | SAGE-217 50 mg (N=268)
Somnolence (Nervous system disorders) | 8 | 41
Dizziness (Nervous system disorders) | 6 | 37
Headache (Nervous system disorders) | 21 | 29
Sedation (Nervous system disorders) | 1 | 20
Nausea (Gastrointestinal disorders) | 12 | 11
Dry Mouth (Gastrointestinal disorders) | 10 | 10
Diarrhoea (Gastrointestinal disorders) | 14 | 8
Tremor (Nervous system disorders) | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT04442490/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT04442490/SAP_001.pdf